CLINICAL TRIAL: NCT03648177
Title: Integrated Psychosocial Group Treatment (IPGT): A Randomized Pilot Trial of a Harm Reduction and Preventative Approach for Patients With Chronic Pain at Risk for Opioid Misuse
Brief Title: Integrative Psychosocial Group Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Staunton Farm Foundation (Unknown)
Responsible Party: Principal Investigator, Valerie Hruschak, PhD Candidate, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO18040067
Record Dates: First submitted 2018-04-04; First posted 2018-08-27 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Chronic Pain; Opioid Misuse
Keywords: Behavioral Intervention; Medication Adherence; Psychosocial Treatment
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Medication Adherence | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Active Comparator: (n=15) Treatment as Usual
  The treatment as usual or control group refers to the standard of care that patients receive for their chronic pain which allows patients to discuss chronic pain with their providers at their discretion. Although highly variable, providers can recommend and prescribe pharmacologic, non-pharmacologic approaches for pain. This study will not interfere in any way with usual care. No additional treatment will be provided to participants allocated to the control group.
  Interventions: Behavioral: Treatment as Usual
- IPGT (Experimental): Experimental: IPGT (n=15) Integrated Psychosocial Group Treatment
  IPGT consists of 6 weekly group sessions of motivational interviewing and behavioral change, self-management, and pain education focused on appropriate adherence to treatment and resisting urges to misuse prescription medications. The intervention also entails an education session on knowledge pertaining to overdose education and naloxone distribution. Topics covered in IPGT include: Pacing and goal setting, negative thinking, coping with stress and anxiety, sleep enhancement techniques, managing set-backs, and chronic pain and your life.
  Interventions: Behavioral: IPGT

INTERVENTIONS:
Behavioral: IPGT — Behavioral Intervention for Patients with Chronic Pain
  Arms: IPGT
Behavioral: Treatment as Usual — Standard Care
  Arms: Treatment as Usual

SUMMARY:
A fundamental challenge for healthcare is to achieve a balance between decreasing the misuse of opioids and associated harms while optimizing patient care, including the provision of multidisciplinary treatments for chronic pain. However, despite recommendations that non-pharmacological interventions are rudimentary in the management of chronic pain, the literature describing which psychosocial interventions are best practice is nearly non-existent. Most of the psychosocial treatments that target either CNCP or opioid misuse are very general and broad-based therapies. However, there is a lack of evidence-informed direction guiding which psychosocial treatments should be adapted to this specialized population and thus, further research is needed.

DETAILED DESCRIPTION:
This project is a pilot randomized controlled trial (RCT) of an Integrated Psychosocial Group Treatment (IPGT) in patients with chronic pain who are at risk for opioid misuse. IPGT is a comprehensive approach that blends evidenced-based psychosocial treatments for chronic pain and opioid misuse and addresses each issue individually, but also the interconnections between the overlapping problems. IPGT consists of 6 weekly group sessions of motivational interviewing and behavioral change, self-management, and pain education focused on appropriate adherence to treatment and resisting urges to misuse prescription medications. The intervention also entails an education session on knowledge pertaining to overdose and naloxone distribution. This study will involve the randomization of 40 patients to receive either: (1) treatment as usual (TAU; n=20); or (2) integrated psychosocial group intervention (IPGT; n=20). This study will: (1) establish feasibility; (2) demonstrate acceptability; and (3) demonstrate preliminary efficacy for an integrated psychosocial group treatment model for patients with chronic pain who are at risk of opioid misuse. The data generated from this study will also serve as a foundation for future implementation to support a subsequent fully-powered RCT.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years)
* chronic pain (3 months or longer)
* at risk for opioid misuse

Exclusion Criteria:

* non-English speaking
* cannot attend group sessions

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of attrition | 12 Months
  Successful delivery of all intervention components to 75% of IPGT recipients.Treatment retention of 75% of IPGT recipients at the completion of the study will be analyzed by calculating number of recipients retained at 6 weeks divided by number of consented recipients.

SECONDARY OUTCOMES:
Acceptability | 12 Months
  Acceptability will be determined with the Patient Satisfaction Questionnaire, a 16 item 5-point Likert scale. All items will be summed up in each subscale and divided by the total number of items to calculate composite scores. The median value of 3.0 will be used as a comparison to determine whether or not the experimental group mean composite scores differ from the hypothesized mean.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Hruschak, PhD Candidate, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Pain Medicine Program, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Hruschak V, Rosen D, Tierney M, Eack SM, Wasan AD, Cochran G. Integrated Psychosocial Group Treatment: A Randomized Pilot Trial of a Harm Reduction and Preventive Approach for Patients with Chronic Pain at Risk of Opioid Misuse. Pain Med. 2021 Sep 8;22(9):2007-2018. doi: 10.1093/pm/pnaa461. PMID 33576415